CLINICAL TRIAL: NCT05947409
Title: Single Arm Clinical Trial of Small Molecule Natural Flavonoid Compounds for Intervention in Neurodegenerative Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mei Han (Other)
Responsible Party: Sponsor-Investigator, Mei Han, Principal Investigator, Beijing University of Chinese Medicine
Organization: Beijing University of Chinese Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMARTO ONE-202305-2
Record Dates: First submitted 2023-06-21; First posted 2023-07-17 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMARTO ONE (Experimental)
  Interventions: Drug: SMARTO ONE

INTERVENTIONS:
Drug: SMARTO ONE — The SMARTO ONE® small molecule natural flavonoid compound product is provided by Beijing Jiafurui Biological Technology Co., Ltd. The intervention agent formula consists of extracts from Polygonum cuspidatum leaves, Fructus ligustri lucidi, Prunus mume, Semen ziziphi spinosae, celery, resistant maltodextrin, and steviol glycoside. Each package of the test product (3g) contains a total flavonoid content of 150mg.

SUMMARY:
1. Explore the effects of natural plant flavonoids on the positive intervention mechanism of neurotransmitter transmission physiological indicators changes (EEG) in the brain of the study subjects;
2. Investigate the effects of natural plant flavonoids in positively intervening clinical symptoms of the study subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 25-70 years
2. Patients complaining of sleep disorders, mood disorders (unstable mood, irritability, depression and anxiety) and cognitive decline (people with memory, decreased reaction time, BPSD symptoms) within one month
3. Montreal Cognitive Assessment Scale (MOCA) score ≤26; if MOCA score is not satisfied, then Pittsburgh Sleep Quality Index (PSQI) score >10 and Hamilton Anxiety Scale (HAMA) score >14 or Hamilton Depression Scale (HAMD) score ≥8 are required
4. Patients who can understand and communicate in language, and complete aphasia patients are not included;
5. Patients who agree to participate in this clinical observation and sign the informed consent form.

Exclusion Criteria:

1. Patients with severe organ diseases such as heart, kidney, and liver failure, chronic lung diseases such as COPD, and severe diabetes;
2. Patients with severe uncontrolled hypertension;
3. Patients who have taken antipsychotic drugs within the past two weeks;
4. Patients with the core features of Lewy body dementia or significant behavioral variant frontotemporal dementia;
5. Patients with various malignant tumors;
6. Patients with progressive stroke, transient ischemic attack, cerebral hemorrhage after cerebral infarction, and cerebral arteritis;
7. Patients with brain tumors, brain trauma, cerebral parasitic diseases, and other conditions;
8. Pregnant or lactating women;
9. Patients allergic to the known ingredients used in this trial;
10. Patients with active ulcers or bleeding tendencies;
11. Patients with neurodegenerative diseases such as Huntington's disease, amyotrophic lateral sclerosis, and Pick's disease;
12. Other patients who are deemed unsuitable to participate in this trial by the investigators.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 4 weeks
  This outcome measure assesses cognitive ability and memory, with evaluation based on a scoring system.The total score ranges from 0 to 30 points, with scores lower than 26 indicating the presence of cognitive impairment. The lower the score, the more severe the disease.
Pittsburgh Sleep Quality Index (PSQI) | 4 weeks
  The evaluation criteria for this outcome measure are as follows: 0-5 points indicate very good sleep quality; 6-10 points indicate average sleep quality; 11-15 points indicate poor sleep quality; 16-21 points indicate very poor sleep quality.
Hamilton Anxiety Rating Scale (HAMA) | 4 weeks
  The evaluation criteria for this outcome measure are as follows: 0-6 points indicate no anxiety symptoms; 7-14 points indicate possible anxiety; 15-21 points indicate definite anxiety; 22-29 points indicate significant anxiety; and scores exceeding 29 points suggest severe anxiety.
Hamilton Depression Scale(HAMD) | 4 weeks
  The evaluation criteria for this outcome measure are as follows:a score of less than 8 is normal, a score of 8-20 may indicate depression, a score of 21-35 may indicate depression, and a score of more than 35 may not indicate severe depression

SECONDARY OUTCOMES:
Numerry of participating with adverse events | baseline, 4 weeks
  This is a safety outcome.
Adverse event occurrence rate | baseline, 4 weeks
  This is a safety outcome.
Abnormality rate of routine blood tests | baseline, 4 weeks
  This is a safety outcome. Included in the outcome indicators are red blood cell count (WBC), haemoglobin concentration (Hb), white blood cell count (WBC), neutrophil count (Neut), lymphocyte count (Lymph), monocyte count (Mono), eosinophil count (Eos), basophil count (Baso) and platelet count (PLT). The abnormal blood count rate was obtained by dividing the number of people with abnormal blood counts by the total number of people with abnormal blood counts.
Liver function-Alanine aminotransferase#ALT# | baseline, 4 weeks
  This is a safety outcome.
Liver function-Aspartate aminotransferase (AST) | baseline, 4 weeks
  This is a safety outcome.
Liver function-Total Protein(TP) | baseline, 4 weeks
  This is a safety outcome.
Electrocardiogram | baseline, 4 weeks
  This is a safety outcome.This outcome measure primarily observes ST segment changes to evaluate the presence or improvement of myocardial ischemia.
Body temperature | baseline, 4 weeks
  This is a safety outcome.
Heart rate | baseline, 4 weeks
  This is a safety outcome.
Number of breaths in 1 min | baseline, 4 weeks
  This is a safety outcome.
Blood pressure-Diastolic blood pressure(mmHg) | baseline, 4 weeks
  This is a safety outcome.
Blood pressure-Systolic blood pressure(mmHg) | baseline, 4 weeks
  This is a safety outcome.